CLINICAL TRIAL: NCT02493478
Title: Observation of Multi-center Quality Improvement Project: Improving Safety and Quality of Tracheal Intubation Practice in Pediatric ICUs
Brief Title: Improving Safety and Quality of Tracheal Intubation Practice in Pediatric ICUs
Acronym: NEAR4KIDs
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 09-007253; R18HS022464 (AHRQ)
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Failed or Difficult Intubation, Sequela; Intubation; Difficult; Intubation Complication
Keywords: Intubation; Advanced airway intervention; Intensive care unit

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Advanced airway interventions are common high risk, high stakes events for children in intensive care units (ICU) and emergency departments (ED), with risk for life and health threatening consequences.

DETAILED DESCRIPTION:
This study will evaluate local pediatric intensive care unit (PICU), cardiac intensive care unit (CICU) and neonatal intensive care unit (NICU) as well as EDs and delivery room (DR) practice, and benchmark against other PICUs, CICUs, NICUs, DRs and EDs as a part of Multi-Center Airway Safety collaborative network (NEAR4KIDS).

The goal of the study is to utilize collected benchmarked data to improve local practice. In order to develop this quality improvement (QI) intervention and collaboration, it is necessary to collect baseline data to describe current practice and to continuously evaluate the effectiveness of any QI intervention.

ELIGIBILITY:
Inclusion Criteria:

* Primary advanced airway events (on patients of all ages) in the PICU, CICU, NICU, DR and ED including: Tracheal Intubation, Laryngeal mask placement, Emergency tracheostomy and/or cricothyrotomy
* Failed extubation attempts or unplanned extubations that require re-intubation will be considered a new primary intubation.

Exclusion Criteria:

* Primary advanced airway events (tracheal intubations, laryngeal mask placement, emergency tracheostomy and/or cricothyrotomy) in the Operating Suites.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All advanced airway events (tracheal intubations, laryngeal mask placement, emergency tracheostomy and cricothyrotomy) in PICUs, CICUs, NICUs, DRs and EDs during study period. Information regarding airway management events as well as select information regarding circumstances up to the event will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2010-03; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of tracheal intubation associated events (TIAEs) | participants will be followed for the duration of their hospital stay, an expected average of 4 weeks
  The number of TIAEs during primary tracheal intubation will be compared to any TIAEs documented during subsequent intubation attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Nadkarni, MD. MS, Principal Investigator — Children's Hospital of Philadelphia
Locations (86):
- United States (63):
  - Children's of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Central California, Madera, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - Nemours Children's Health, Delaware, Wilmington, Delaware
  - Miami Children's Hospital, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Children's Hospital of Atlanta - Scottish Rite, Atlanta, Georgia
  - Children's Hospital of Georgia, Augusta, Georgia
  - Northwestern Medicine Prentice Women's Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Beacon Children's Hospital, South Bend, Indiana
  - Kentucky Children's Hospital, Lexington, Kentucky
  - Norton Children's Hospital - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Medicine, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Gillette Children's Specialty Health, Saint Paul, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - Children's Hospital and Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Albany Medical College, Albany, New York
  - Oishei Children's Hospital, Buffalo, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - New York Presbyterian Hospital Weill Cornell Medical College, New York, New York
  - University of Rochester at Golisano Children's Hospital, Rochester, New York
  - Stony Brook Children's Hospital, Stony Brook, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Maria Fareri Children's Hospital (West Chester Medical), Valhalla, New York
  - Duke Children's Hospital, Durham, North Carolina
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital - Penn State Hershey, Hershey, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Dell Children's Medical Center - Ascension, Austin, Texas
  - Medical City Children's Hospital, Dallas, Texas
  - Baylor - Christus Children's - Main Hospital, Irving, Texas
  - Baylor - Christus Children's - Westover Hills, San Antonio, Texas
  - Baylor - Christus Children's - Stone Oak, San Antonio, Texas
  - The University of Vermont Children's Hospital, Burlington, Vermont
  - UVA Children's Hospital, Charlottesville, Virginia
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin - UnityPoint Meriter, Madison, Wisconsin
  - American Family Children's Hospital - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - University of Wisconsin - American Family Children's Hospital, Shorewood Hills, Wisconsin
- Australia (2):
  - Royal Brisbane and Women's Hospital, Herston
  - The Royal Children's Hospital Melbourne, Parkville
- Medical University of Vienna (Medizinische Universität Wien), Vienna, Austria
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CHU Sainte-Justine, Montreal, Quebec
  - The University of Manitoba, Winnipeg
- University Hospital Schleswig-Holstein, Campus Luebeck, Children's Hospital, Lübeck, Germany
- India (2):
  - Aster Hospitals - India, Bengaluru, Karnataka
  - Rainbow Children's Hospital, Bangalore
- Bambino Gesu, Roma, Italy
- Japan (7):
  - National Center for Child Health and Development, Setagaya-Ku, Tokyo
  - Hiroshima University, Hiroshima
  - Hyogo Prefectural Kobe Children's Hospital, Kobe
  - Aichi Children's Health and Medical Center, Ōbu
  - Saitama Children's Medical Center, Saitama
  - Jichi Medical University Hospital, Shimotsuke
  - Tokyo Metropolitan, Tokyo
- Starship Children's Hospital, Auckland, New Zealand
- Singapore (2):
  - KK Women's and Children's Hospital, Singapore
  - KK Women's & Children's Hospital, Singapore, Singapore
- Cardiff & Vale University Health Board, Cardiff, Wales, United Kingdom

REFERENCES:
- [Derived] Gabrani A, Kojima T, Sanders RC Jr, Shenoi A, Montgomery V, Parsons SJ, Gangadharan S, Nett S, Napolitano N, Tarquinio K, Simon DW, Lee A, Emeriaud G, Adu-Darko M, Giuliano JS Jr, Meyer K, Graciano AL, Turner DA, Krawiec C, Bakar AM, Polikoff LA, Parker M, Harwayne-Gidansky I, Crulli B, Vanderford P, Breuer RK, Gradidge E, Branca A, Glater-Welt LB, Tellez D, Wright LV, Pinto M, Nadkarni V, Nishisaki A; National Emergency Airway Registry for Children (NEAR4KIDS) Collaborators and Pediatric Acute Lung Injury and Sepsis Investigators (PALISI). Downward Trend in Pediatric Resident Laryngoscopy Participation in PICUs. Pediatr Crit Care Med. 2018 May;19(5):e242-e250. doi: 10.1097/PCC.0000000000001470. PMID 29406378